CLINICAL TRIAL: NCT00686946
Title: The National Register of Antipsychotic Medication in Pregnancy (NRAMP)
Acronym: NRAMP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Alfred (Other)
Collaborators: Janssen-Cilag Ltd. (Industry); AstraZeneca (Industry); Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Jayashri Kulkarni, Professor, Chief Investigator, The Alfred
Other Study IDs: 114/04
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy; Mental Disorders
Keywords: Severe mental illness; Antipsychotic medications; Pregnancy; Evidence-based guidelines; Maternal and infant health and wellbeing
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NRAMP: Participants take their antipsychotic medication as prescribed by their clinical treating teams.

SUMMARY:
The National Register of Antipsychotic Medication in Pregnancy (NRAMP)is an observational, nationwide study involving women of child-bearing age who take antipsychotic medication during pregnancy. It follows the pathway of mother and baby during pregnancy and for the first 12 months of the baby's life, in order to develop evidence-based guidelines for the best use and effect of antipsychotic medication during pregnancy, thereby informing clinical treating teams with regard to the management of their patients in this vulnerable population group.

The investigators hypothesize that the provision of such evidence-based guidelines will improve the management and outcomes for mother and baby during pregnancy, birth and the postnatal phase, providing a positive impact on maternal and child health and wellbeing for present and future generations.

DETAILED DESCRIPTION:
The desire to reproduce is both a powerful urge and a basic human right for women regardless of mental health status. Deinstitutionalised treatment for mental illness, better pharmacotherapies, and generally higher expectations for a normal quality of life have the potential to raise the incidence of pregnancy in women with psychosis (Miller, Bloom & Resnick, 1992). The right of women with mental illness to become parents places responsibility upon health care professionals to ensure sound antenatal and ongoing care is available.

Ethical duty of care aside, good antenatal treatment appears prudent given the greater risk of obstetric complications in women with schizophrenia (Sacker et al, 1996). In a meta analysis of studies examining outcomes for pregnant women with and without schizophrenia, evidence exists of a small but statistically significant increase in the risk of low birth weight and inferior neonatal condition in infants of the schizophrenia cohort (Sacker et al, 1996). A recent meta analysis (Webb, et al, 2005) summarized that exposure to maternal psychotic illness is associated with a "higher than expected" risk of perinatal and infant mortality, including an almost twofold chance of fetal death or stillbirth (p.1052). Jablensky and colleagues (2005) further discovered that women whose psychiatric illness commenced before the birth of their child were significantly more likely to experience obstetric complications than women whose first admission for mental illness was after the delivery. Moreover, the offspring of women with schizophrenia carry with them an increased risk for developing psychosis (Mednick, Parnas & Schulsinger, 1987). This observation has driven the neurodevelopmental hypothesis about the aetiology of schizophrenia, which posits that alterations to early fetal brain development in utero might lead to a predisposition to the formation of schizophrenia later in life (Lewis & Murray, 1987). Such perinatal contributions to adult mental health outcomes points to the necessity to provide pregnant women who have psychosis, with proper and specialized treatment.

Despite these clear arguments for a thorough understanding of the needs of pregnant women with schizophrenia, current research is limited. In particular, there is currently very little evidence regarding the use of antipsychotic medication in pregnancy upon fetal development and maternal health. Over the last four decades, intermittent studies have sought to investigate the teratogenicity of the older or typical antipsychotics upon fetal development. Earlier reports were generated from pregnancy outcomes of women treated with these medications for hyperemesis gravidarum, not from women with schizophrenia (Kerns, 1989); as such, it is difficult to extrapolate initial findings across these two cohorts with confidence. Limb defects in children born to women who were given large doses of haloperidol in early pregnancy are outlined in case reports (Goldberg & Nissam, 1994). Patton and colleagues (2002) also reviewed three other larger studies and concluded that a significant increased chance exists for babies exposed to phenothiazines to develop congenital malformations, compared with the incidence within the general population.

The newer or second generation antipsychotics (SGAs) have not been studied in any great detail; to date, to our knowledge, there have been no blinded or randomized studies examining birth outcomes in women taking SGAs, and these are unlikely given ethical considerations. Prescribing guidelines laid out in MIMS (2003) for all current SGAs include pregnancy as a "special precaution" and despite the gravity of associated risks of teratogenesis, there are few publications examining atypical antipsychotic medication use in pregnant women. In their review, Patton and colleagues (2002) cite four studies on the outcome of clozapine use, noting that for a total five cases no congenital abnormalities were reported, although one infant experienced low grade fever and seizure, with gastroesophageal reflux. Grigoriadis and Seeman (2002) suggest that the increased risk of agranulocytosis and seizures in babies, coupled with the identification of both pregnancy and clozapine as potentially increasing the likelihood of thromboembolisms, render this a medication to be avoided during pregnancy. Twenty-three Olanzapine-exposed pregnancies were observed by Goldstein and colleagues (2000), who found there was no increased risk of spontaneous abortion, stillbirth, prematurity or major malformation. The authors were, however, swift to assert that studies of greater sample sizes and over a protracted time period are necessary before olanzapine can be declared "safe" with confidence.

Thus, clinicians remain in a conundrum; although in general today's antipsychotic drugs produce fewer side effects, are better tolerated by the patient, and more effectively target the symptoms of psychosis, little evidence has been presented to reassure prescribers that their impact upon fetal development is minimal. A proven, evidence based method for achieving a balance between maternal mental health with minimal risk to the fetus must be researched and evidenced. Therefore, we have established The National Register of Antipsychotic Medication in Pregnancy (NRAMP) as a non-interventional means of providing information about pregnancies and outcomes for women with psychosis, and their babies. Not only is NRAMP seeking to record large scale obstetric information in a prospective fashion, including pharmacotherapy during pregnancy and beyond, it is also capitalizing on the opportunity to track alterations to mental health symptoms of women during pregnancy and in the post partum period, and to gather valuable insights into the attitudes of this cohort as they make the transition into parenthood.

The combination of poor psychosocial history, existing involvement with child protection agencies, psychiatric diagnoses and admissions, medications and substance abuse, present many issues affecting outcomes for both mother and child during the perinatal period. Our study involves extensive collaboration between many different clinical groups, and will culminate in an important best-practice resource to improve the quality of life for both present and future generations. The identification of a history of serious mental illness and a planned management strategy are therefore essential if we are to improve outcomes for mother and baby.

This then, is the driving force behind the establishment of The National Register of Antipsychotic Medication in Pregnancy (NRAMP), and is a much-needed strategy to improve the management of serious mental illness for women who become pregnant.

This investigator initiated study has been funded by Janssen-Cilag, AstraZeneca, Hospira, Lilly and the Australian Rotary Health Research Fund. NB: AstraZeneca provided funding up to and including 250 consented participants. The study continues to recruit.

ELIGIBILITY:
Inclusion Criteria:

* Women who take antipsychotic medication during pregnancy
* Women who are pregnant or have had a baby in the last 12 months
* Women who are living in Australia
* Women who are able to provide informed consent

Exclusion Criteria:

* Women who do not take antipsychotic medication during pregnancy
* Women who are not pregnant, or have not had a baby in the last 12 months
* Women who are unable to provide informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women from across Australia who are taking, or have taken, antipsychotic medication during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2005-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Participant interviews | Antenatal - once per trimester; Postnatal - quarterly for 12 months
  Interviews to gather demographic, social, medical, psychiatric, medication and obstetric history

SECONDARY OUTCOMES:
Psychopathology measures for the mother | Antenatal and up to 12 months postnatally
  PANSS (Positive and Negative Syndrome Scale) Questionnaire EPDS (Edinburgh Postnatal Depression Scale)Questionnaire
Developmental Milestone measures for the baby | Birth to 12 months of age
  ASQ-3 (Ages and Stages Questionnaire, Third Edition)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Jayashri Kulkarni, MBBS,FRANZCP, Principal Investigator — Monash Alfred Psychiatry Research Centre (MAPrc)
Locations (1):
- Monash Alfred Pyschiatry Research Centre, Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared, for example, in Case Studies, where personal identification is not compromised, which also allows for an aggregate view of data.